CLINICAL TRIAL: NCT04173871
Title: Effects of Systematic Proprioceptive-tactile Stimulation With Use of the Protac MyFit®
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Protac A/S (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RoTilFokus_USouthernDenmark
Record Dates: First submitted 2019-10-31; First posted 2019-11-22 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Sensory Processing Disorder; Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group
  Interventions: Device: Protac Myfit®
- Control (No Intervention): Control group

INTERVENTIONS:
Device: Protac Myfit® — A systematic proprioceptive-tactile stimulation by the Protac MyFit® vest. The children are asked to wear the Protac Myfit® vest from the beginning of every school day and for at least two sessions for three weeks.
  Arms: Intervention

SUMMARY:
Children with sensory impairment (SPD) are often unable to sit still and focus their attention. This can affect the children by limiting their opportunities for participation in school activities. Previous studies indicate a link between childhood SPD, childhood anxiety, and obsessive-compulsive disorder (OCD) in adulthood. Research and clinical experience suggest that systematic use of proprioceptive-tactile stimulant aids may have a positive effect for children with SPD.

The aim of the project is to investigate and describe the effects of a systematic use of proprioceptive-tactile stimulating vest, MyFit®, for children 6-12 years with SPD in the form of sensory-seeking behaviour.

Research questions:

* Can systematic use of MyFit® for children with sensory seeking behaviour increase their participation in school activities?
* Can systematic use of MyFit® support children with sensory seeking behaviour to increase their awareness, concentration and focus on tasks?
* Can systematic use of MyFit® affect children's feelings of confidence and self-efficacy? The project seeks to answer these questions to contribute to knowledge on how children with sensory seeking behaviours can be supported for better participation in school activities.

The study will be a randomized controlled trial of 240 children with SPD and sensory seeking behaviour.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the effect of systematic proprioceptive-tactile stimulation through use of the Protac MyFit® to children, age 6-12 years with SPD and sensory seeking behavior. The primary objective is to determine the effect of the vest on the children´s abilities for attention and participation in school activities, and secondary their abilities for on-task behavior and feelings of self-esteem and self-efficacy.

Method & design The study is a randomized controlled trial (RCT), were primary school children with SPD and sensory seeking behavior receives an intervention with systematic proprioceptive-tactile stimulation through use of the Protac MyFit®.

Study setting and participants The study will be conducted in public primary schools across Denmark. Participants will be 240 children with SPD and sensory seeking behaviour age 6-12 years attending public primary school. Sample size has been calculated based on results from the feasibility study and the primary outcome of sustained attention measured with the Test of Every Day Attention-Children. The sample size is calculated with Ancova analysis and made with an anticipated difference on 1.5 with a correlation of .07 and a standard deviation at 5.

Recruitment and randomization Recruitment will be conducted in collaboration with gatekeepers from municipal Pedagogical Psychological Counselling (PPR) departments and public-school managements across Denmark, that will assist in identifying possible study participants. Parents to possible participants will be introduced to the study by the gatekeepers and handed out written information about the study together with a baseline questionnaire, the Short Sensory Profile questionnaire (SSP), a consent form for participation and a franked reply envelope.

The included children will be randomized into two groups; an intervention group (A) and a control group (B). The randomization will be computer generated 1:1. Additionally, 20 of the included children will be strategically selected (as per age, gender, group) to represent the main population and complete a qualitative research interview regarding their experiences of using the MyFit®.

Intervention The intervention consisted of systematic proprioceptive-tactile stimulation by the MyFit®, were the children are asked to wear the vest from the beginning of every school day within the study period. Additionally, the participants are invited to use the vest as they please at home and doing leisure activities.

At baseline participants try out and chose whether they wish to use a vest with balls 25mm or 38mm in diameter. Doing the test period participants in both group A and B will receive the usual treatment as provided by the PPR departments, the school and/or the family doctor. Usual treatment offered by PPR and schools can vary between municipalities, it can be in form of physical therapy, occupational therapy, increased support doing school activities etc. This will be registered and described throughout the study. Parents of participant are asked to document if the child receive any other treatment medical or otherwise.

Participation in the study will be voluntary and the families will be informed that they at any time can withdraw from the study and that the child should never be forced to use the vest.

ELIGIBILITY:
Inclusion Criteria:

* Children age 6-12 years, with SPD and sensory seeking behaviour as identified by the SSP, attending primary school.

Exclusion Criteria:

* Children with mental retardation or other massive cognitive impairment, and children who use corset or molded wheelchairs.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Test of Everyday Attention - Children (TEA-Ch) | 21 days
  TEA-Ch is a normed and standardised battery of 9 tests, that examines the child's ability for three different types of attention (selective attention, sustained attention and attentional control/switching)
Child Occupational Self Assessment (COSA) | 21 days
  COSA is an assessment tool designed to capture children´s perceptions of their own occupational competence together with their rating of importance of everyday activities.

SECONDARY OUTCOMES:
Registration of on-task-behaviour | 21 days
  Study specifik registration tool.
Five to fifteen (FTF) | 21 days
  A standardized questionnaire to parents, that gives an overview of a child's neuropsychological and behavioural function and examine the child´s development in different areas (181 items in total). In this study we have included the domain regarding executive functions and the subdomain of body perception in a questionnaire to the parents. Additionally, we have included the domain regarding learning in a questionnaire to the teachers.
Strengths and Difficulties Questionnaire (SDQ) | 21 days
  A standardized questionnaire to teachers and parents, that screen for positive and negative psychological attributes in children age 3 - 16 years. In this study we only use the SDQ to the teachers and only the 13 items regarding school activities and social behaviour.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Natasja Nielsen, PhD. Student, Principal Investigator — University of Southern Denmark
Locations (1):
- National Institute of Public Health, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No